CLINICAL TRIAL: NCT01597622
Title: BEL114333, a Multicenter, Continuation Study of Belimumab in Subjects With Systemic Lupus Erythematosus (SLE) Who Completed the Phase III Study BEL113750 in Northeast Asia or Completed the Open-label Extension of HGS1006-C1115 in Japan
Brief Title: BEL114333, a Continuation Study of BEL113750 in Subjects With Systemic Lupus Erythematosus (SLE) in Northeast Asia, and in Japan Subjects Completing the Open-label Extension of HGS1006-C1115
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Human Genome Sciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 114333
Record Dates: First submitted 2012-05-10; First posted 2012-05-14 (Estimated); Results first posted 2020-01-09 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Systemic Lupus Erythematosus
Keywords: SELENA; belimumab; Lupus; systemic lupus erythematosus; PGA; BLys; SLE Flare Index; continuation; phase III; BILAG; extension; efficacy; SRI; B cell; SLEDAI; safety; Asia; B lymphocyte
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — belimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open-label Belimumab (Experimental): Belimumab 10 mg/kg administered intravenously every 4 weeks. All study subjects will receive standard SLE therapies during the study. Subjects will continue to receive belimumab treatment until such time belimumab becomes commercially available in a subject's country of participation, or the subject elects to participate in another belimumab continuation study for SLE, or until either the subject's physician withdraws the subject from the study, or upon the decision by the sponsor to discontinue further development of belimumab for SLE.
  Interventions: Drug: Belimumab

INTERVENTIONS:
Drug: Belimumab — 10 mg/kg administered intravenously over 1 hour every 4 weeks

SUMMARY:
This study provides subjects who complete the BEL113750 study and subjects who complete the open-label extension of HGS1006-C1115 (referred to as C1115) Study in Japan the option of continuing treatment with belimumab (10 mg/kg intravenously every 4 weeks) for those randomized to belimumab, or the option to begin treatment with belimumab for those randomized to placebo, as an add-on to their standard of care SLE therapy.

DETAILED DESCRIPTION:
This is a multicentre, continuation study of belimumab plus standard of care (SOC) in SLE subjects who completed the Phase III BEL113750 protocol in Northeast Asia or who completed the open-label extension of the HGS1006-C1115 protocol in Japan. This study provides subjects who complete the BEL113750 study the option of continuing treatment with belimumab (10 mg/kg intravenously every 4 weeks) for those randomized to belimumab, or the option to begin treatment with belimumab for those randomized to placebo, as an add-on to their SOC SLE therapy. Subjects participating in this continuation protocol will continue to be monitored for safety and efficacy, as measured by the SLE responder index. Subjects who complete 48 weeks of treatment on the BEL113750 study and who meet inclusion/exclusion criteria, and provide informed consent, will be given the option to enter the continuation study. All subjects will receive belimumab 10 mg/kg IV infused over 1 hour every 4 weeks. Subjects recruited into this study will continue to receive treatment with belimumab until such time as belimumab becomes commercially available in a subject's country of participation, or the subject elects to participate in another belimumab continuation study for SLE, or until either the subject's physician withdraws the subject from the study, or upon the decision by the sponsor to discontinue further development of belimumab for SLE.

ELIGIBILITY:
Inclusion Criteria:

* Have completed the BEL113750 Protocol in Northeast Asia through Week 48 OR have completed the open-label extension of C1115 in Japan.
* Be able to receive the first dose of belimumab for BEL114333 four weeks (minimum of 2 weeks, maximum of 8 weeks) after the last dose in BEL113750 OR be able to receive the first dose of IV belimumab 1 week (plus a 1 week visit window) after the last dose of open-label SC belimumab in C1115..

Exclusion Criteria:

* Have developed clinical evidence of significant, unstable or uncontrolled, acute or chronic diseases not due to SLE (i.e., cardiovascular, pulmonary, hematologic, gastrointestinal, hepatic, renal, neurological, malignancy or infectious diseases), or experienced an adverse event (AE) in the Phase 3 study that could, in the opinion of the principal investigator, put the subject at undue risk.
* Have developed any other medical diseases (e.g., cardiopulmonary), laboratory abnormalities, or conditions (e.g., poor venous access) that in the opinion of the principal investigator, makes the subject unstable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2012-06-11 (Actual); Primary Completion 2018-09-13 (Actual); Study Completion 2018-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (17):
- Japan (12):
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Ehime
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Hiroshima
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Miyagi
  - GSK Investigational Site, Nagasaki
  - GSK Investigational Site, Okayama
  - GSK Investigational Site, Okinawa
  - GSK Investigational Site, Tochigi
  - GSK Investigational Site, Tokyo
- South Korea (5):
  - GSK Investigational Site, Busan
  - GSK Investigational Site, Daegu
  - GSK Investigational Site, Incheon
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Suwon, Kyonggi-do

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20307

REFERENCES:
- [Derived] Tanaka Y, Bae SC, Bass D, Curtis P, Chu M, DeRose K, Ji B, Kurrasch R, Lowe J, Meizlik P, Roth DA. Long-term open-label continuation study of the safety and efficacy of belimumab for up to 7 years in patients with systemic lupus erythematosus from Japan and South Korea. RMD Open. 2021 Jul;7(2):e001629. doi: 10.1136/rmdopen-2021-001629. PMID 34215703

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was multicenter, open-label continuation study of belimumab plus standard of care (SOC) in Systemic Lupus Erythematosus (SLE) participants who completed study BEL113750 (NCT01345253) in Northeast Asia (Japan and Korea) & participants who completed the open-label extension of C1115 (NCT01484496) in Japan to assess long term safety & efficacy.
Pre-assignment Details: Total 143 participants were screened for this study and 142 participants were enrolled and received study treatment in current study. BEL113750, a 52 week double-blind study; C1115, a 52 week double-blind study followed by a 6 month open-label extension.
Groups:
- Open-label Belimumab 10 mg/kg: Participants received Belimumab 10 milligrams (mg)/kilogram (kg) intravenously (IV) over 1 hour on Week 0, Week 4 and then every 4 weeks until Week 48 of the first year (Study Year 1); on Week 4 and then every 4 weeks until Week 48 of subsequent years during study (up to Study Year 7 Week 4 Visit, which represents a maximum duration of 5 years and 7 months by calendar year in this open-label study. One Study Year is 48 weeks). All participants were continued on their SOC therapies as prescribed by the investigator.
Period: Overall Study
Arm/Group | Open-label Belimumab 10 mg/kg
Started | 142
Completed | 104
Not Completed | 38
Not completed — Adverse Event | 7
Not completed — Lack of Efficacy | 3
Not completed — Protocol Violation | 1
Not completed — Lost to Follow-up | 1
Not completed — Investigator Discretion | 5
Not completed — Withdrawal by Subject | 20
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: Baseline is the last available value prior to the first belimumab exposure.
Groups:
- Open-label Belimumab 10 mg/kg: Participants received Belimumab 10 milligrams (mg)/kilogram (kg) intravenously (IV) over 1 hour on Week 0, Week 4 and then every 4 weeks until Week 48 of the first year (Study Year 1); on Week 4 and then every 4 weeks until Week 48 of subsequent years during study (up to Study Year 7 Week 4 Visit, which represents a maximum duration of 5 years and 7 months by calendar year in this open-label study. One Study Year is 48 weeks). All participants were continued on their SOC therapies as prescribed by the investigator. First belimumab exposure is the first dose in parent study, for participant randomized to belimumab in the parent study; and first OL belimumab dose received (i.e. in either C1115 open-label extension, or BEL114333), for participant randomized to placebo in parent study.
Arm/Group | Open-label Belimumab 10 mg/kg
Number analyzed (Participants) | 142
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.6 (9.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 129
  Male | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaskan Native | 1
  Japanese Heritage | 71
  East Asian Heritage | 68
  Southeast Asian Heritage | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious AEs (SAEs)
Description: Any untoward medical occurrence in participant, temporally associated with use of medicinal product, whether or not considered related to medicinal product. Any untoward event resulting in death,life threatening,requires hospitalization or prolongation of existing hospitalization,results in disability/incapacity,congenital anomaly/birth defect,medically important were categorized as SAE. Number of participants who had any AE(includes those having non-serious and/or serious AEs) or any SAE are presented.Treatment-emergent AEs are defined as AEs that started on or after first dose of belimumab treatment and for those participants who were randomized to placebo in parent study,ongoing AEs that started before first open-label belimumab dose(in either C1115 open-label extension or BEL114333),worsened (severity,seriousness,relatedness) at any point during the open-label treatment.Timeframe includes exposure in parent study/upto16 weeks post infusion in current study(114333).
Time Frame: Up to 6 calendar years and 9 months
Population: Safety Population. All participants in the Enrolled population who received at least one IV dose of belimumab during current study.
Measure: Count of Participants; unit: Participants
Arm/Group | Open-label Belimumab 10 mg/kg
Number analyzed (Participants) | 142
Participants
  Any SAEs | 48
  Any AEs | 139

2. Secondary Outcome: Percentage of SLE Responder Index (SRI) Responders by Study Visit
Description: SRI response is composite index, defined as percent of participants with>=4 point reduction from Baseline in safety of estrogen in lupus national assessment systemic lupus erythematosus disease activity index (SELENA-SLEDAI) score and no worsening (increase of <0.30 points from Baseline) in physicians global assessment(PGA) &no new British isles lupus assessment group (BILAG) A organ domain score or 2 new BILAG B organ domain scores compared with Baseline at the time of assessment. A SELENA SLEDAI score of 0 would suggest no lupus activity; while a score of 105 is the maximum calculable if all items were scored as being present from active lupus. PGA ranges from 0(no activity) to 3(severe activity). BILAG has no range. Baseline is last available value prior to first belimumab exposure. Year 8 Week 24 visit is the Exit Visit obtained by slotting the Exit Visit to Week 24. Timeframe includes exposure in parent study/upto 4 weeks post infusion (Exit visit) in current study (114333).
Time Frame: Study Years 1 to 7: At Week 24 and 48 Visits, Year 8: only Week 24 Visit
Population: Safety Population. Only those participants with data available at the specified data points were analyzed (represented by n=X in the category title)
Measure: Number; unit: Percentage of Participants
Arm/Group | Open-label Belimumab 10 mg/kg
Number analyzed (Participants) | 142
Percentage of Participants
  Year 1 Week 24, n=136: number analyzed (Participants) | 136
  Year 1 Week 24, n=136 | 47.8
  Year 1, Week 48, n=133: number analyzed (Participants) | 133
  Year 1, Week 48, n=133 | 51.1
  Year 2, Week 24, n=129: number analyzed (Participants) | 129
  Year 2, Week 24, n=129 | 55.0
  Year 2, Week 48, n=121: number analyzed (Participants) | 121
  Year 2, Week 48, n=121 | 53.7
  Year 3, Week 24, n=103: number analyzed (Participants) | 103
  Year 3, Week 24, n=103 | 57.3
  Year 3, Week 48, n=88: number analyzed (Participants) | 88
  Year 3, Week 48, n=88 | 68.2
  Year 4, Week 24, n=80: number analyzed (Participants) | 80
  Year 4, Week 24, n=80 | 67.5
  Year 4, Week 48, n=60: number analyzed (Participants) | 60
  Year 4, Week 48, n=60 | 76.7
  Year 5, Week 24, n=32: number analyzed (Participants) | 32
  Year 5, Week 24, n=32 | 71.9
  Year 5, Week 48, n=29: number analyzed (Participants) | 29
  Year 5, Week 48, n=29 | 69.0
  Year 6, Week 24, n=24: number analyzed (Participants) | 24
  Year 6, Week 24, n=24 | 66.7
  Year 6, Week 48, n=22: number analyzed (Participants) | 22
  Year 6, Week 48, n=22 | 68.2
  Year 7, Week 24, n=18: number analyzed (Participants) | 18
  Year 7, Week 24, n=18 | 83.3
  Year 7, Week 48, n=13: number analyzed (Participants) | 13
  Year 7, Week 48, n=13 | 84.6
  Year 8, Week 24, n=1: number analyzed (Participants) | 1
  Year 8, Week 24, n=1 | 100

ADVERSE EVENTS:
Time Frame: Treatment-emergent SAEs and non-serious AEs were collected up to maximum duration of 6 calendar years and 9 months.
Description: Treatment-emergent SAEs and non-serious AEs were reported for the Safety Population consisted of all participants in the enrolled population who received at least one IV dose of belimumab during current study. Timeframe includes exposure in parent study/up to 16 weeks post infusion of treatment in current study 114333.
Arm/Group | Open-label Belimumab 10 mg/kg
All-Cause Mortality (participants affected / at risk) | 1/142
Serious Adverse Events (participants affected / at risk) | 48/142
Other Adverse Events (participants affected / at risk) | 134/142
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-label Belimumab 10 mg/kg (N=142)
Cellulitis (Infections and infestations) | 3 (3)
Herpes zoster (Infections and infestations) | 3 (3)
Endocarditis (Infections and infestations) | 2 (2)
Pyelonephritis acute (Infections and infestations) | 2 (2)
Abscess jaw (Infections and infestations) | 1 (1)
Atypical pneumonia (Infections and infestations) | 1 (1)
Bacterial pyelonephritis (Infections and infestations) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 1 (1)
External ear cellulitis (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Gastroenteritis salmonella (Infections and infestations) | 1 (1)
Genital herpes zoster (Infections and infestations) | 1 (1)
Herpes dermatitis (Infections and infestations) | 1 (1)
Herpes simplex pharyngitis (Infections and infestations) | 1 (1)
Infectious colitis (Infections and infestations) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1)
Pelvic inflammatory disease (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (2)
Pneumonia bacterial (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1)
Tuberculous pleurisy (Infections and infestations) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 3 (3)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 1 (2)
Lupus pancreatitis (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 2 (2)
Oedema peripheral (General disorders) | 1 (3)
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Cutaneous lupus erythematosus (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Systemic lupus erythematosus rash (Skin and subcutaneous tissue disorders) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Protein urine present (Investigations) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 2 (2)
Brain stem infarction (Nervous system disorders) | 1 (1)
Putamen haemorrhage (Nervous system disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 1 (2)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pericarditis lupus (Cardiac disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Diabetes insipidus (Endocrine disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Open-label Belimumab 10 mg/kg (N=142)
Nasopharyngitis (Infections and infestations) | 86
Viral upper respiratory tract infection (Infections and infestations) | 25
Herpes zoster (Infections and infestations) | 23
Upper respiratory tract infection (Infections and infestations) | 22
Influenza (Infections and infestations) | 20
Gastroenteritis (Infections and infestations) | 18
Pharyngitis (Infections and infestations) | 14
Bronchitis (Infections and infestations) | 13
Cystitis (Infections and infestations) | 12
Oral herpes (Infections and infestations) | 11
Urinary tract infection bacterial (Infections and infestations) | 11
Hordeolum (Infections and infestations) | 9
Conjunctivitis (Infections and infestations) | 8
Abdominal pain upper (Gastrointestinal disorders) | 23
Nausea (Gastrointestinal disorders) | 23
Diarrhoea (Gastrointestinal disorders) | 22
Constipation (Gastrointestinal disorders) | 17
Abdominal pain (Gastrointestinal disorders) | 16
Vomiting (Gastrointestinal disorders) | 16
Dental caries (Gastrointestinal disorders) | 13
Dyspepsia (Gastrointestinal disorders) | 11
Dermatitis contact (Skin and subcutaneous tissue disorders) | 13
Rash (Skin and subcutaneous tissue disorders) | 12
Eczema (Skin and subcutaneous tissue disorders) | 10
Acne (Skin and subcutaneous tissue disorders) | 9
Urticaria (Skin and subcutaneous tissue disorders) | 9
Back pain (Musculoskeletal and connective tissue disorders) | 18
Arthralgia (Musculoskeletal and connective tissue disorders) | 16
Myalgia (Musculoskeletal and connective tissue disorders) | 16
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11
Headache (Nervous system disorders) | 40
Dizziness (Nervous system disorders) | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 26
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 10
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 9
Contusion (Injury, poisoning and procedural complications) | 16
Ligament sprain (Injury, poisoning and procedural complications) | 11
Thermal burn (Injury, poisoning and procedural complications) | 8
Pyrexia (General disorders) | 19
Oedema peripheral (General disorders) | 11
Insomnia (Psychiatric disorders) | 17
Dysmenorrhoea (Reproductive system and breast disorders) | 8
Hypertension (Vascular disorders) | 11
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8
Vertigo (Ear and labyrinth disorders) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-05-31): https://cdn.clinicaltrials.gov/large-docs/22/NCT01597622/SAP_000.pdf
  • Study Protocol (2014-05-16): https://cdn.clinicaltrials.gov/large-docs/22/NCT01597622/Prot_001.pdf